CLINICAL TRIAL: NCT05895383
Title: Self-Adjusted Nitrous Oxide: A Feasibility Study in the Setting of Vasectomy
Acronym: SANO-VAS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Heidi Rayala, Assistant Professor of Surgery, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023P-000328
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Procedural Pain; Pain Catastrophizing; Procedural Anxiety
Keywords: vasectomy; nitrous oxide; experience of care; ambulatory
MeSH Terms: conditions — Pain, Procedural | interventions — Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: All participants will receive nitrous oxide at levels of mild sedation during vasectomy. Participants will hold a remote control to adjust the level of gas administered according to their comfort level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Self-adjusted nitrous oxide (SANO) (Experimental): All patients will receive nitrous oxide at concentrations of minimal sedation (0-50%) throughout vasectomy.
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: Nitrous oxide — Nitrous oxide administered at concentrations of minimal sedation (0-50%). Participants will be able to adjust the level of gas throughout the vasectomy using a handheld remote control.
  Other Names: Self-adjusted nitrous oxide

SUMMARY:
This study is being done to see if nitrous oxide during vasectomy decreases pain and anxiety, and also assess whether patients have better satisfaction when they control their own level of nitrous oxide during the procedure. If we find that patients experience less pain or anxiety with nitrous oxide, it could be suggested that self-adjusted nitrous oxide (SANO) may be a useful tool for improving experience of care during vasectomy.

DETAILED DESCRIPTION:
Patients scheduled for vasectomy at Beth Israel Deaconess Medical Center will be contacted and offered enrollment in the study. Vasectomy will occur according to standard-of-care and all participants will receive the typical lidocaine injections at the beginning of the procedure. Before the start of the vasectomy, a study staff member will help participants put on a plastic gas mask and demonstrate how to turn the gas up or down using the remote control. Nitrous oxide and oxygen will be given through a plastic mask. A remote control given to participants will allow them to adjust the nitrous oxide based on their comfort. The Nitrouseal® machine used in this study limits nitrous oxide to concentrations to "minimal sedation" (0-50%), which are levels where a person remains awake and is able to talk and breath normally.

Before the day of a participant's vasectomy, they will be asked questions related to demographics and medical history to determine study eligibility. Immediately before and after vasectomy, participants will be asked to describe their anxiety and pain levels. At two-weeks and three-months after vasectomy, a brief electronic survey will be sent to participants' email asking about recollection of pain and anxiety and satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for vasectomy
2. Aged 21 to 85 years
3. Suitable for receipt of inhaled nitrous oxide/oxygen
4. Access to an email and computer

Exclusion Criteria:

1. Perioral facial hair impeding good mask seal
2. Cognitive impairment that impedes ability to complete survey questions
3. Intent to use benzodiazepines or opioids "as needed" for purposes of vasectomy
4. Has any of the following medical conditions, which contraindicate use of nitrous oxide:

   1. Inner ear, bariatric or eye surgery within the last 2 weeks,
   2. Current emphysematous blebs,
   3. Severe B-12 deficiency,
   4. Bleomycin chemotherapy within the past year,
   5. Heart attack within the past year,
   6. Stroke within the past year,
   7. Class III or higher heart failure.

Ages: 21 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Procedural pain assessed by the Visual Analog Scale for Pain (VAS-P) | Measured immediately after completion of vasectomy
  Level of pain experienced during vasectomy as measured by the Visual Analog Scale for Pain (VAS-P; range: 0 no pain - 10 worst pain).

SECONDARY OUTCOMES:
Anticipated pain assessed by the Visual Analog Scale for Pain (VAS-P) | Measured immediately prior to vasectomy
  Level of anxiety anticipated during vasectomy as measured by the Visual Analog Scale for Pain (VAS-P; range: 0 no pain - 10 worst pain).
Anticipated anxiety assessed by the Visual Analog Scale for Anxiety (VAS-A) | Measured immediately prior to vasectomy
  Level of anxiety anticipated during vasectomy as measured by the Visual Analog Scale for Anxiety (VAS-A; range: 0 no anxiety - 10 worst anxiety).
Procedural anxiety assessed by the Visual Analog Scale for Anxiety (VAS-A) | Measured immediately after completion of vasectomy
  Level of anxiety experienced during vasectomy as measured by the Visual Analog Scale for Anxiety (VAS-A; range: 0 no anxiety - 10 worst anxiety).
Recalled pain assessed by the Visual Analog Scale for Pain (VAS-P) | Measured two weeks and three months after vasectomy
  Level of pain recalled during vasectomy as measured by the Visual Analog Scale for Pain (VAS-P; range: 0 no pain - 10 worst pain).
Recalled anxiety assessed by the Visual Analog Scale for Pain (VAS-P) | Measured two weeks and three months after vasectomy
  Level of anxiety recalled during vasectomy as measured by the Visual Analog Scale for Anxiety (VAS-A; range: 0 no anxiety - 10 worst anxiety).
Satisfaction assessed by Likert scale | Measured during and two weeks after vasectomy
  Satisfaction of concentration of SANO during vasectomy will be measured by the maximum concentration of SANO reached during the procedure compared to participants' response to: "How do you feel about the level of SANO you received during the vasectomy?" (less than I would like, about right, more than I would like) and "How helpful do you think SANO was in relieving your pain and anxiety?" (very helpful, unhelpful, undecided, helpful very helpful).
Operator ease of performing vasectomy | Measured immediately after urologist finishes vasectomy
  Operating urologist will be asked to fill out a three-item "operator survey" that asks if "Patient tolerated lidocaine injection," "Patient maintained positioning," and "Patient tolerated vasectomy," "Worse than expected (-1)", "As expected (0)" or "Better than expected (+1)." The composite score will be used as a measure of operator ease.
Emergent adverse events as assessed by frequency of incidents | Measured during and up to 30 days after day of vasectomy
  Emergent adverse events possibly related to SANO will be recorded by frequency on the day-of the vasectomy and by monitoring participants' online medical record up to 30 days after the vasectomy. Termination of SANO during the vasectomy due to discomfort, nausea, or vomiting will also be considered as adverse events related to SANO.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Rayala, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center; Marissa Kent, MD, Study Chair — Beth Israel Deaconess Medical Center; Peter Steinberg, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No